CLINICAL TRIAL: NCT04360889
Title: Lipid Peroxidation and Options Antioxidant Therapy for Secondary Lymphedema of the Lower Extremities
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ryazan State Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MDA-1
Record Dates: First submitted 2020-04-18; First posted 2020-04-24 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Lower Extremity Lymphedema
Keywords: endothelial dysfunction; secondary lymphedema of the lower extremities; antioxidants; micronized purified flavonoid fraction
MeSH Terms: interventions — Hesperidin; Tocopherols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Tocopherol (Experimental): patients with lower limb lymphedema who will receive conservative therapy with elastic compression and an antioxidant (Tocopherol-400 IU/day) - 90 days
  Interventions: Drug: Tocopherol
- Micronised purified flavonoid fraction (Experimental): patients with lower limb lymphedema who will receive conservative therapy with Micronised purified flavonoid fraction (diosmin+flavonoids expressed as hesperidin)-1000mg/day) in addition to elastic compression - 90 days
  Interventions: Drug: Micronised purified flavonoid fraction (diosmin+flavonoids expressed as hesperidin)
- Elastic compression (Other): patients with lower limb lymphedema who will be treated with elastic compression - 90 days
  Interventions: Other: Elastic compression
- Healthy volunteers (No Intervention): healthy volunteers with no history or clinical signs of venous or lymphatic disease - 90 days

INTERVENTIONS:
Drug: Micronised purified flavonoid fraction (diosmin+flavonoids expressed as hesperidin) — Micronised purified flavonoid fraction (diosmin+flavonoids expressed as hesperidin) is prescribed at a dose of 1000 mg / day Tocopherol is prescribed at a dose of 400 ME/ day
  Arms: Micronised purified flavonoid fraction
Drug: Tocopherol — patients with lower limb lymphedema receiving conservative therapy (elastic compression, to which are added preparations with antioxidant endotheliotropic activity (Tocopherol-400 IU/day)
  Arms: Tocopherol
Other: Elastic compression — patients with lower limb lymphedema receiving conservative therapy that includes only the use of elastic compression
  Arms: Elastic compression

SUMMARY:
A single-center, open, prospective, randomized, controlled clinical trial will include 120 patients with lower limb lymphedema who undergo treatment in an office-based vascular lab at the Ryazan regional clinical cardiology dispensary, Ryazan, Russia. The patients will be recruited by the staff of the Department of cardiovascular, endovascular, operative surgery, and topographic anatomy, Ryazan state I.P. Pavlov medical university, Russia. The study will include patients who meet the inclusion criteria and do not meet the exclusion criteria. Patients will be divided into 4 groups, 30 subjects each. Group 1-patients with lower limb lymphedema who will receive conservative therapy with elastic compression and an antioxidant (Tocopherol-400 IU/day); Group 2-patients with lower limb lymphedema who will receive conservative therapy with Micronised purified flavonoid fraction (diosmin+flavonoids expressed as hesperidin)-1000mg/day) in addition to elastic compression; Group 3-patients with lower limb lymphedema who will be treated with elastic compression; Group 4- healthy volunteers with no history or clinical signs of venous or lymphatic disease; The duration of this study for each subject will be a maximum of 90 days. Pre-screening and screening will involve 200 subjects with a total of 120 subjects who will be randomized into the study. Peripheral blood samples will be collected to evaluate the activity of biochemical markers of endothelial function; the quality of life will also be assessed.

DETAILED DESCRIPTION:
Research methods:

1. Physical examination;
2. peripheral blood sampling (assessment of the concentration of the markers of endothelial dysfunction, including malondialdehyde (MDA), superoxide dismutase (SD), catalase( CAT), glutathione peroxidase (GP). MDA concentration will be determined with a competitive enzyme immunoassay (ELISA), which will be performed using a General MDA assessment kit (manufacturer: USCN Life Science Inc. US-CEA597GE). CAT concentration will be determined using a competitive enzyme immunoassay (ELISA), which will be performed with a kit for quantitative in vitro assessment of catalase (manufacturer: USCN Life Science Inc. US-SEC418Hu). GP concentration will be determined with a competitive enzyme immunoassay (ELISA), which will be performed using a glutathione peroxidase quantification set (abfrontier supplier, Republic of Korea - LF- EK0110). SOD concentration will be determined using a competitive enzyme immunoassay (ELISA), which will be performed using a total superoxide dismutase detection kit (supplier Cayman Chemical Company, US - 706002).
3. Lower limb venous sonography with a linear 5-13 MHz probe;
4. Patient questionnaire using a Russian-language version of the Quality of life questionnaire "SF-36 Health Status Survey"

ELIGIBILITY:
Inclusion Criteria:

* Secondary lymphedema of the lower extremities
* Signed Informed Consent Form

Exclusion Criteria:

* varicose veins of the lower extremities,
* deep vein thrombosis,
* post-thrombotic disease,
* obliterating
* atherosclerosis of the lower limb arteries,
* pregnancy,
* lactation,
* cancer,
* acute violation of cerebral circulation in the anamnesis,
* trophic lesions of the skin of the lower extremities,
* diabetes mellitus
* an infectious disease with a history of three months prior to inclusion in the study,
* heart failure,
* kidney failure,
* pulmonary insufficiency.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-08-03 (Actual); Study Completion 2022-08-03 (Actual)

PRIMARY OUTCOMES:
The malleolar volume of the limb | 90 days
  The circumference at the level of the narrowest part of the lower leg, measured in centimeters
The Level Of Catalase | 90 days
  Biochemical indicator of the functional state of the endothelium. Catalase concentration will be determined using a competitive enzyme immunoassay (ELISA), which will be performed with a kit for quantitative in vitro assessment of catalase (manufacturer: USCN Life Science Inc. US-SEC418Hu). Unit of measurement ng / ml
The Level Of Superoxide Dismutase | 90 days
  Biochemical indicator of the functional state of the endothelium. Superoxide Dismutase concentration will be determined using a competitive enzyme immunoassay (ELISA), which will be performed using a total superoxide dismutase detection kit (supplier Cayman Chemical Company, US - 706002). Unit of measurement UI / ml
The Level Of Glutathione Peroxidase | 90 days
  Biochemical indicator of the functional state of the endothelium. Glutathione Peroxidase concentration will be determined with a competitive enzyme immunoassay (ELISA), which will be performed using a glutathione peroxidase quantification set (abfrontier supplier, Republic of Korea - LF- EK0110). Unit of measurement ng / ml
The level of Malondialdehyde | 90 days
  Biochemical indicator of the functional state of the endothelium. Malondialdehyde concentration will be determined with a competitive enzyme immunoassay (ELISA), which will be performed using a General MDA assessment kit (manufacturer: USCN Life Science Inc. US-CEA597GE). Unit of measurement ng / ml
Quality of life indicators: questionnaire | 90 days
  Patient questionnaire using a Russian-language version of the Quality of life questionnaire "Short Form-36 Health Status Survey". 8 indicators. Indicator from 0 to 100. Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Ryazan State Medical University, Ryazan, Russia

IPD SHARING:
Plan to Share IPD: No